CLINICAL TRIAL: NCT01781663
Title: Efficacy of KAM2904 Face Cream and KAM3008 Body Lotion Treatment in Children With Atopic Dermatitis (AD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kamedis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAM-ATOPIC-01
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KAM2904 Face Cream and KAM3008 Body Lotion (Experimental): A group treated with KAM2904 Face Cream and KAM3008 Body Lotion
  Interventions: Device: KAM2904 Face Cream; Device: KAM3008 Body Lotion
- petrolatum-based moisturizer (Sham Comparator): control group
  Interventions: Other: petrolatum-based moisturizer

INTERVENTIONS:
Device: KAM2904 Face Cream
  Arms: KAM2904 Face Cream and KAM3008 Body Lotion
Device: KAM3008 Body Lotion
  Arms: KAM2904 Face Cream and KAM3008 Body Lotion
Other: petrolatum-based moisturizer
  Arms: petrolatum-based moisturizer

SUMMARY:
The main purpose of this study is to demonstrate the safety and efficacy of KAM2904 Face Cream and KAM3008 Body Lotion in reducing the symptoms of mild to moderate AD. Efficacy will be evaluated by comparing SCORAD and Eczema Area Severity Index (EASI) in a group of subjects treated with KAM2904 Face Cream and KAM3008 Body Lotion (the treatment group), versus a group of subjects treated with a petrolatum-based moisturizer (the control group). Safety will be determined by the number and severity of Adverse Events Device-Related.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female between 2 and 12 years of age

  * The subject suffers from moderate atopic dermatitis (SCORAD<40) that is amenable to treatment
  * Diagnosis of atopic dermatitis meets Hanifin's criteria (at least 3 basic features and at least 3 minor features)
  * Atopic dermatitis is, in the opinion of the investigator, stable for the past 7 days
  * The subject's parents are able to apply the study product twice a day (each morning and evening) for a consecutive period of 42 days
  * The subject's parents agree that the subject will not change his/her lifestyle during the study period (including: regular body hygiene product (soap), the number of baths and showers per day, the laundry detergent and fabric softener used to wash clothes)
  * The subject's parents agree to use only the test product during the study period
  * The subject's legal guardian is able and willing to sign the informed consent form and to comply with the study regulations of this protocol

Exclusion Criteria:

* • The subject has another dermatological disease/condition that could interfere with the clinical evaluation, including infected atopic dermatitis lesions

  * The subject has a previous history of allergy to cosmetic products or to any of the ingredients included in the tested formulations (Appendices 1 and 2)
  * The subject received a topical or a systemic immune-modulator (such calcineurin inhibitors or cortico-steroids) for the treatment of atopic dermatitis, within 14 days prior to day 0
  * The subject underwent phototherapy within 28 days prior to day 0
  * The subject is expected to be extensively exposed to the sun during the trial
  * The subject underwent any experimental treatment within 14 days prior to day 0

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
• Change in SCORAD (Scoring Atopic Dermatitis) | after 42 days of treatment
• Change in EASI (Eczema Area Severity Index) | after 42 days of treatment
• Change in the scoring of individual symptoms of atopic dermatitis | after 42 days of treatment

SECONDARY OUTCOMES:
• Trend in the change of SCORAD | after 42 days of treatment
• Trend in the change of EASI | after 42 days of treatment
• Trend in the change of individual symptoms of atopic dermatitis | after 42 days of treatment
• Safety of KAM2904 Face Cream and KAM3008 Body Lotion | days D14, D28, D42 and unscheduled visits
  Safety will be measured by the number and severity of Device-Related Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eli Sprecher, MD, Principal Investigator — Tel Aviv Soraski Medical Center - Dermatology Unit
Locations (1):
- Fundación Teknon, Barcelona, Spain

REFERENCES:
- See also: Sponsor's site — http://www.kamedis.com